CLINICAL TRIAL: NCT03271489
Title: A Phase 3b Study to Evaluate the Long-Term Safety of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: Long-Term Safety Study of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-283
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Heavy Menstrual Bleeding; Uterine Fibroids
Keywords: Elagolix Sodium; Heavy Menstrual Bleeding (HMB); Heavy Uterine Bleeding; Leiomyomata; Menorrhagia; Elagolix + Norethindrone Acetate; Elagolix + E2/NETA; Elagolix; Safety; Efficacy
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — elagolix; Estradiol; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elagolix plus estradiol (E2)/norethindrone acetate (NETA) (Experimental)
  Interventions: Drug: Elagolix; Drug: Estradiol /norethindrone acetate (E2/NETA)
- Placebo (Placebo Comparator)
  Interventions: Other: E2/NETA Placebo; Other: Elagolix Placebo

INTERVENTIONS:
Drug: Elagolix — Film-coated 300 mg tablets
  Arms: Elagolix plus estradiol (E2)/norethindrone acetate (NETA)
Drug: Estradiol /norethindrone acetate (E2/NETA) — Estradiol 1 mg/norethindrone acetate 0.5 mg capsules
  Arms: Elagolix plus estradiol (E2)/norethindrone acetate (NETA)
Other: E2/NETA Placebo — Placebo capsules
  Arms: Placebo
Other: Elagolix Placebo — Film-coated placebo tablets
  Arms: Placebo

SUMMARY:
This randomized multicenter phase 3b study seeks to evaluate the safety of elagolix in combination with estradiol/norethindrone acetate for the management of heavy menstrual bleeding associated with uterine fibroids in premenopausal women. This study was double-blind (DB) during the first 12 months and open-label (OL) for the next 36 months.

DETAILED DESCRIPTION:
478 participants were randomly assigned at a ratio of 2:1 to the following treatment groups:

1. Elagolix 300 mg twice daily (BID) plus estradiol 1.0 mg/norethindrone acetate 0.5 mg (E2/NETA) once daily (QD) for 48 months, followed by 12 months PTFU
2. Placebo for 12 months, followed by elagolix 300 mg BID plus E2/NETA QD for 36 months, followed by 12 months PTFU

This study was double-blinded during the first 12 months and open-label for the next 36 months. Participants entered up to 12 months of PTFU after completing treatment Month 48 (or at any time a participant prematurely discontinued treatment).

ELIGIBILITY:
Inclusion Criteria:

* Participant is a premenopausal female at the time of Screening.
* Participant has a diagnosis of uterine fibroids documented by a Pelvic Ultrasound [Transabdominal ultrasound (TAU) or transvaginal ultrasound (TVU)].
* Participant has Heavy Menstrual Bleeding (HMB) associated with uterine fibroids as evidenced by Menstrual Blood Loss (MBL) > 80 mL during each of two screening menses as measured by the alkaline hematin method.
* Participant has negative urine and/or serum pregnancy test during Washout (if applicable) and/or Screening and just prior to first dose.
* Participant has an adequate endometrial biopsy performed during Screening, the results of which show no clinical significant endometrial pathology.

Exclusion Criteria:

* Participant has screening pelvic ultrasound or Saline Infusion Sonohysterography (SIS) results that show a clinically significant gynecological disorder.
* Participant has history of osteoporosis or other metabolic bone disease.
* Participant has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis.
* Participant has a history of major depression or post-traumatic stress disorder (PTSD) episode within 2 years of screening, OR a history of other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder).
* Participant is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over the counter and prescription topical, inhaled, intranasal or intra-articular injectable (for occasional use) corticosteroids are allowed.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 478 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (157):
- United States (155):
  - Alabama Clinical Therapeutics /ID# 160835, Birmingham, Alabama
  - Alabama Clinical Therapeutics /ID# 160927, Birmingham, Alabama
  - Choice Research, LLC /ID# 161498, Dothan, Alabama
  - Southern Women's Specialists PC /ID# 161531, Fairhope, Alabama
  - E Squared Research /ID# 163645, Huntsville, Alabama
  - Women's Health Alliance of Mobile /ID# 161443, Mobile, Alabama
  - Mobile, OBGYN P.C. /ID# 161530, Mobile, Alabama
  - Mesa Obstetricians and Gynecologists /ID# 160955, Mesa, Arizona
  - Noble Clinical Research /ID# 166949, Tucson, Arizona
  - Vision's Clinical Research-Tucson /ID# 161508, Tucson, Arizona
  - Eclipse Clinical Research /ID# 161516, Tucson, Arizona
  - Duplicate_Core Healthcare Group /ID# 160858, Cerritos, California
  - Diagnamics Inc. /ID# 160950, Encinitas, California
  - HRC Fertility /ID# 161493, Encino, California
  - SC Clinical Research /ID# 164395, Garden Grove, California
  - Duplicate_Duplicate_Marvel Clinical Research /ID# 167297, Huntington Beach, California
  - Grossmont Ctr Clin Research /ID# 165120, La Mesa, California
  - Olympia Clinical Trials /ID# 201562, Los Angeles, California
  - National Research Institute /ID# 160952, Los Angeles, California
  - Futura Research, Org /ID# 160924, Montebello, California
  - California Medical Research Associates /ID# 161481, Northridge, California
  - Northern California Research /ID# 161561, Sacramento, California
  - Precision Research Institute - San Diego /ID# 163069, San Diego, California
  - MD Strategies Research Centers /ID# 161544, San Diego, California
  - Health care Affiliates Medical Group /ID# 163324, Santa Ana, California
  - Alta California Medical Group /ID# 163564, Simi Valley, California
  - Upland Clinical Research /ID# 164528, Upland, California
  - Bayview Research Group LLC /ID# 161484, Valley Village, California
  - Advanced RX Clinical Research /ID# 161599, Westminster, California
  - Emerson Clinical Research Inst /ID# 162181, Washington D.C., District of Columbia
  - James A. Simon, MD, PC /ID# 160931, Washington D.C., District of Columbia
  - Women's Health Partners /ID# 203577, Boca Raton, Florida
  - David Lubetkin MD LLC /ID# 203578, Boca Raton, Florida
  - Brandon Premier Health Care, PA/Gulf Coast Research Group, LLC /ID# 160910, Brandon, Florida
  - Omega Research Maitland, LLC /ID# 160857, DeBary, Florida
  - Midland Florida Clinical Research Center /ID# 161487, DeLand, Florida
  - KO Clinical Research, LLC /ID# 160928, Fort Lauderdale, Florida
  - Sweet Hope Research Specialty Inc /ID# 163522, Hialeah, Florida
  - Solutions Through Adv Rch /ID# 160935, Jacksonville, Florida
  - Altus Research, Inc /ID# 160912, Lake Worth, Florida
  - Wellington Anti-Aging Centre /ID# 203540, Loxahatchee Groves, Florida
  - South Florida Wellness & Clinic /ID# 161535, Margate, Florida
  - Invictus Clinical Research Group,LLC /ID# 160925, Miami, Florida
  - Healthcare Clinical Data, Inc /ID# 160888, Miami, Florida
  - Palmetto Professional Research /ID# 161442, Miami, Florida
  - Vista Health Research, LLC /ID# 163044, Miami, Florida
  - Duplicate_Precision Research Organization /ID# 161522, Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc /ID# 161549, Miami Springs, Florida
  - Salom Tangir, LLC /ID# 162542, Miramar, Florida
  - Advanced Research Institute, Inc /ID# 163748, New Port Richey, Florida
  - A Premier Medical Research of FL /ID# 201882, Orange City, Florida
  - Clinical Associates of Orlando /ID# 160889, Orlando, Florida
  - Oncova Clinical Research, Inc. /ID# 160937, Saint Cloud, Florida
  - Physician Care Clin. Res., LLC /ID# 161547, Sarasota, Florida
  - Accel Research Sites - St Petersburg Clinical Research Unit /ID# 160913, St. Petersburg, Florida
  - Treasure Coast Research /ID# 161824, Stuart, Florida
  - Discovery Clinical Research /ID# 160891, Sunrise, Florida
  - Precision Clinical Research /ID# 165377, Sunrise, Florida
  - GCP Clinical Research, LLC /ID# 164593, Tampa, Florida
  - University of South Florida- Neuroscience Institute /ID# 160960, Tampa, Florida
  - Jedidiah Clinical Research /ID# 167114, Tampa, Florida
  - Virtus Research Consultants, LLC /ID# 160855, Wellington, Florida
  - Comprehensive Clinical Trials LLC /ID# 161479, West Palm Beach, Florida
  - Journey Medical Research Insti /ID# 160958, Alpharetta, Georgia
  - Paramount Research Solutions /ID# 161557, Alpharetta, Georgia
  - AGILE Clinical Research Trials /ID# 160941, Atlanta, Georgia
  - Mount Vernon Clinical Res, LLC /ID# 161491, Atlanta, Georgia
  - Atlanta Women's Research Institute /ID# 160844, Atlanta, Georgia
  - Medisense Inc /ID# 161494, Atlanta, Georgia
  - Duplicate_Atlanta Gynecology Research Institute /ID# 160851, Suwanee, Georgia
  - Bingham Memorial Hospital /ID# 201130, Blackfoot, Idaho
  - Leavitt Womens Healthcare /ID# 163419, Idaho Falls, Idaho
  - Womens Healthcare Assoc, DBA /ID# 160933, Idaho Falls, Idaho
  - Sonora Clinical Research /ID# 167610, Meridian, Idaho
  - Asr, Llc /Id# 162179, Nampa, Idaho
  - Women's Health Practice, LLC /ID# 161553, Champaign, Illinois
  - Moore for Women Healthcare and Wellness Institute, LLC /ID# 167118, Chicago, Illinois
  - Duplicate_University of Chicago /ID# 162667, Chicago, Illinois
  - Alliance for Multispecialty Research, LLC /ID# 160932, Oak Brook, Illinois
  - Women's Health Advantage /ID# 161537, Fort Wayne, Indiana
  - Womens & Family Care, LLC dba /ID# 160890, Shawnee Mission, Kansas
  - Bluegrass Clinical Research /ID# 163485, Louisville, Kentucky
  - Clinical Trials Management, LLC - Covington /ID# 160838, Covington, Louisiana
  - Clinical Trials Management, LLC - Covington /ID# 160893, Covington, Louisiana
  - Praetorian Pharmaceutical Research /ID# 161532, Marrero, Louisiana
  - Ochsner Baptist Medical Centre /ID# 161507, New Orleans, Louisiana
  - Women Under Study, LLC /ID# 163990, New Orleans, Louisiana
  - Willis-Knighton Pediatric GI S /ID# 161534, Shreveport, Louisiana
  - Exordia Medical Research, Inc /ID# 160853, Fall River, Massachusetts
  - Duplicate_Great Lakes Research Group, Inc. /ID# 161511, Bay City, Michigan
  - Wayne State University /ID# 160944, Detroit, Michigan
  - Valley OB-Gyn Clinic - Saginaw /ID# 203579, Saginaw, Michigan
  - Saginaw Valley Med Res Group /ID# 160840, Saginaw, Michigan
  - Quad Clinical Research, LLC /ID# 200943, St Louis, Missouri
  - Excel Clinical Research /ID# 165588, Las Vegas, Nevada
  - Office of Edmond E. Pack, MD /ID# 162604, Las Vegas, Nevada
  - Private practice: Dr. Rex G. Mabey JR /ID# 160915, Las Vegas, Nevada
  - Jersey Shore University Medical Center /ID# 160916, Neptune City, New Jersey
  - Lovelace Scientific Resources /ID# 163644, Albuquerque, New Mexico
  - Bosque Women's Care /ID# 162606, Albuquerque, New Mexico
  - SUNY Downstate Medical Center /ID# 160922, Brooklyn, New York
  - Duplicate_Northwell Health System - Manhasset /ID# 201058, Manhasset, New York
  - Columbia Univ Medical Center /ID# 161519, New York, New York
  - Hamburg Regional Gynecology Gr /ID# 161427, Orchard Park, New York
  - DJL Clinical Research, PLLC /ID# 161548, Charlotte, North Carolina
  - Carolina Women's Research and Wellness Center /ID# 160914, Durham, North Carolina
  - Unified Women's Clinical Resea /ID# 163014, Raleigh, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 161490, Raleigh, North Carolina
  - Unified Women's Clinical Resea /ID# 160957, Winston-Salem, North Carolina
  - Clinical Inquest Center Ltd /ID# 160892, Beavercreek, Ohio
  - Duplicate_CTI Clinical Research Center /ID# 160942, Cincinnati, Ohio
  - Univ Hosp Cleveland /ID# 160953, Cleveland, Ohio
  - Central Ohio Clinical Research /ID# 201162, Columbus, Ohio
  - Duplicate_Optimed Research /ID# 165600, Columbus, Ohio
  - Hilltop Obstetrics & Gynecology /ID# 203576, Middletown, Ohio
  - University of Toledo /ID# 160923, Toledo, Ohio
  - Oregon Medical Research Center /ID# 161514, Portland, Oregon
  - OB/GYN Associates of Erie /ID# 161541, Erie, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 160896, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 160936, Philadelphia, Pennsylvania
  - DUP_Thomas Jefferson University /ID# 200304, Philadelphia, Pennsylvania
  - Vista Clinical Research /ID# 160946, Columbia, South Carolina
  - VitaLink Research-Spartanburg /ID# 164592, Spartanburg, South Carolina
  - Duplicate_Chattanooga Medical Research /ID# 160885, Chattanooga, Tennessee
  - WR-ClinSearch /ID# 160887, Chattanooga, Tennessee
  - The Jackson Clinic, PA /ID# 162496, Jackson, Tennessee
  - Research Memphis Associates, LLC /ID# 160939, Memphis, Tennessee
  - OBGYN North /ID# 203580, Austin, Texas
  - Austin Area Obstetrics, Gynecology, and Fertility /Id# 203542, Austin, Texas
  - Discovery Clinical Trials -HCWC /ID# 161543, Dallas, Texas
  - Duplicate_The University of Texas Southwestern Medical Center /ID# 161496, Dallas, Texas
  - Baylor Scott & White /ID# 161515, Fort Worth, Texas
  - Willowbend Health and Wellness - Frisco /ID# 160954, Frisco, Texas
  - The Ob/Gyn Center /ID# 165928, Houston, Texas
  - Precision Research Institute, LLC /ID# 161554, Houston, Texas
  - The Woman's Hospital of Texas /ID# 160959, Houston, Texas
  - Centex Studies, Inc /ID# 163858, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 160917, Houston, Texas
  - UAG Innovation Women Research, /ID# 167415, Houston, Texas
  - America's Adv. Wellness Center /ID# 167548, Houston, Texas
  - FMC Science /ID# 160886, Lampasas, Texas
  - Advances in Health, Inc. /ID# 160930, Pearland, Texas
  - ClinRx Research, LLC /ID# 201170, Plano, Texas
  - Clinical Trials of Texas, Inc /ID# 161510, San Antonio, Texas
  - VIP Trials /ID# 161546, San Antonio, Texas
  - Houston Ctr for Clin Research /ID# 160837, Sugar Land, Texas
  - The Univ Texas HSC at Tyler /ID# 161533, Tyler, Texas
  - Center of Reproductive Medicine /ID# 162498, Webster, Texas
  - Univ of Virgnia Medical center /ID# 166283, Charlottesville, Virginia
  - Eastern Virginia Med School /ID# 160856, Norfolk, Virginia
  - Clinical Research Partners /ID# 160929, North Chesterfield, Virginia
  - Clinical Research Partners /ID# 160948, North Chesterfield, Virginia
  - Clinical Trials Virginia, Inc. /ID# 160943, Richmond, Virginia
  - Specialists for Women /ID# 201129, Suffolk, Virginia
  - Tidewater Clinical Research /ID# 160949, Virginia Beach, Virginia
- Puerto Rico (2):
  - Henry A. Rodriguez Ginorio, MD /ID# 160861, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 160862, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 478 participants were enrolled across the United States and Puerto Rico.
Groups:
- Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA): Participants were randomized to receive elagolix 300 mg BID plus E2/NETA (estradiol 1 mg/norethindrone acetate 0.5 mg QD) for 48 months followed by 12 months post-treatment follow-up
- Placebo: Participants were randomized to receive placebo for 12 months, followed by elagolix 300 mg BID plus E2/NETA (estradiol 1 mg/norethindrone acetate 0.5 mg QD) for 36 months followed by 12 months post-treatment follow-up
Period: Screening Period
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Started | 319 | 159
Completed | 319 | 159
Not Completed | 0 | 0
Period: Double-Blind (DB) Period
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Started | 319 | 159
Completed | 283 | 135
Not Completed | 36 | 24
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Lost to Follow-up | 9 | 9
Not completed — Requires surgery or invasive intervention for treatment of uterine fibroids | 3 | 2
Not completed — Non-compliance with study procedures | 0 | 1
Not completed — Other | 6 | 1
Not completed — Missing | 1 | 0
Period: Open-Label (OL) Period
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Started | 193 | 84
Completed | 159 | 68
Not Completed | 34 | 16
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Lost to Follow-up | 10 | 5
Not completed — Non-compliance with study procedures | 4 | 1
Not completed — No Specified | 2 | 2
Not completed — Missing | 2 | 0
Period: Post-Treatment Follow-Up (PTFU) Period
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Started | 319 | 159
Completed | 189 | 86
Not Completed | 130 | 73
Not completed — Adverse Event | 16 | 6
Not completed — Withdrawal by Subject | 40 | 26
Not completed — Lost to Follow-up | 35 | 24
Not completed — Requires surgery or invasive intervention for treatment of uterine fibroids | 5 | 3
Not completed — Non-compliance with study procedures | 9 | 2
Not completed — COVID-19 logistical restrictions | 1 | 0
Not completed — Other | 21 | 10
Not completed — Missing | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo | Total
Number analyzed (Participants) | 319 | 159 | 478
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (5.07) | 41.7 (5.65) | 42.3 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 159 | 478
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 31 | 108
  Not Hispanic or Latino | 242 | 128 | 370
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 171 | 99 | 270
  White | 128 | 51 | 179
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
  AEs during the 12-month DB period were defined as any AEs with onset on/after first dose of study drug during the DB period and no more than 30 days after the last dose of study drug for participants who discontinued early during the DB period, or until the first dose of study drug in the OL period for participants who entered the OL Treatment Period. AEs during the OL period were defined as AEs with onset on/after first dose of study drug during the OL period and no more than 30 days after the last dose of study drug. During the post-treatment follow-up (PTFU) period, adverse events were collected from 30 days post-last dose until end of study. Safety reporting during the PTFU period included AESIs. Other AEs may have also been reported.
Time Frame: Baseline to 60 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Number analyzed (Participants) | 319 | 159
Participants
  Double-blind Period | 203 | 83
  Open-label Period: number analyzed (Participants) | 193 | 84
  Open-label Period | 124 | 59
  Post-treatment Follow-up Period | 22 | 6

2. Secondary Outcome: Bone Mineral Density (BMD) Recovery After up to 48 Months of Treatment
Description: Percent Recovery of BMD after 6 and 12 months of post-treatment follow-up (PTFU) for Spine, Total Hip, and Femoral Neck. BMD assessments were measured by dual X-ray absorptiometry (DXA). Analysis excludes participants who switched machine manufacturer type. Percent recovery is defined as 100*(% change from Baseline to final on-treatment assessment - % change from Baseline to post-treatment visit) / (% change from Baseline to final on treatment assessment) and is defined only for subjects with BMD decrease at final on-treatment assessment.
Time Frame: Baseline through Month 60
Population: Of the total participants in the Safety Analysis Set, each row includes participants with a BMD decrease from baseline at their final on-treatment visit (up to Month 48), in any location (spine, total hip or femoral neck), and at least 1 DXA scan during the follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Elagolix Plus Estradiol (E2)/Norethindrone Acetate (NETA) | Placebo
Number analyzed (Participants) | 111 | 40
Participants
  Spine (6 months PTFU): number analyzed (Participants) | 54 | 19
  Spine (6 months PTFU): < 0% Recovery | 24 | 10
  Spine (6 months PTFU): 0% - 25% Recovery | 8 | 2
  Spine (6 months PTFU): > 25% - 50% Recovery | 3 | 2
  Spine (6 months PTFU): > 50% - 75% Recovery | 5 | 2
  Spine (6 months PTFU): > 75% - 100% Recovery | 5 | 1
  Spine (6 months PTFU): > 100% Recovery | 9 | 2
  Spine (12 months PTFU): number analyzed (Participants) | 65 | 22
  Spine (12 months PTFU): < 0% Recovery | 23 | 10
  Spine (12 months PTFU): 0% - 25% Recovery | 3 | 2
  Spine (12 months PTFU): > 25% - 50% Recovery | 5 | 1
  Spine (12 months PTFU): > 50% - 75% Recovery | 9 | 2
  Spine (12 months PTFU): > 75% - 100% Recovery | 5 | 0
  Spine (12 months PTFU): > 100% Recovery | 20 | 7
  Total Hip (6 months PTFU): number analyzed (Participants) | 51 | 17
  Total Hip (6 months PTFU): < 0% Recovery | 20 | 10
  Total Hip (6 months PTFU): 0% - 25% Recovery | 5 | 1
  Total Hip (6 months PTFU): > 25% - 50% Recovery | 5 | 4
  Total Hip (6 months PTFU): > 50% - 75% Recovery | 7 | 1
  Total Hip (6 months PTFU): > 75% - 100% Recovery | 1 | 0
  Total Hip (6 months PTFU): > 100% Recovery | 13 | 1
  Total Hip (12 months PTFU): number analyzed (Participants) | 66 | 19
  Total Hip (12 months PTFU): < 0% Recovery | 22 | 12
  Total Hip (12 months PTFU): 0% - 25% Recovery | 11 | 1
  Total Hip (12 months PTFU): > 25% - 50% Recovery | 7 | 1
  Total Hip (12 months PTFU): > 50% - 75% Recovery | 6 | 2
  Total Hip (12 months PTFU): > 75% - 100% Recovery | 5 | 0
  Total Hip (12 months PTFU): > 100% Recovery | 15 | 3
  Femoral Neck (6 months PTFU): number analyzed (Participants) | 51 | 20
  Femoral Neck (6 months PTFU): < 0% Recovery | 22 | 10
  Femoral Neck (6 months PTFU): 0% - 25% Recovery | 5 | 2
  Femoral Neck (6 months PTFU): > 25% - 50% Recovery | 8 | 1
  Femoral Neck (6 months PTFU): > 50% - 75% Recovery | 5 | 4
  Femoral Neck (6 months PTFU): > 75% - 100% Recovery | 4 | 1
  Femoral Neck (6 months PTFU): > 100% Recovery | 7 | 2
  Femoral Neck (12 months PTFU): number analyzed (Participants) | 60 | 22
  Femoral Neck (12 months PTFU): < 0% Recovery | 18 | 10
  Femoral Neck (12 months PTFU): 0% - 25% Recovery | 12 | 2
  Femoral Neck (12 months PTFU): > 25% - 50% Recovery | 7 | 1
  Femoral Neck (12 months PTFU): > 50% - 75% Recovery | 6 | 3
  Femoral Neck (12 months PTFU): > 75% - 100% Recovery | 3 | 1
  Femoral Neck (12 months PTFU): > 100% Recovery | 14 | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from time of informed consent to the end of the study. The median time participants were followed for the screening period was: 106 days (PBO) and 113 days (ELA/E2-NETA); double blind period: 335 days (PBO) and 336 days (ELA/E2-NETA); open label period: 555 days (PBO to ELA/E2-NETA) and 681 days (ELA/E2-NETA to ELA/E2-NETA); long-term follow-up period: 197 days (PBO to ELA/E2-NETA) and 324 days (ELA/E2-NETA to ELA/E2-NETA).
Description: Safety reporting during the PTFU period included Adverse Events of Special Interest (AESIs). Other AEs may have also been reported.
Groups:
- Screening Placebo: AEs and SAEs during the screening period were collected from the time of informed consent to the first dose of placebo (approximately 2.5 to 5 months).
- Screening Elagolix E2/NETA: AEs and SAEs during the screening period were collected from the time of informed consent to the first dose of Elagolix E2/NETA (approximately 2.5 to 5 months).
- Double-Blind Placebo: Participants received 12 months of treatment with placebo. AEs and SAEs during the Double-Blind treatment period were collected from the first dose of placebo to the start of the open label period (12 months).
- Double-Blind Elagolix E2/NETA: Participants received 12 months of treatment with elagolix 300 mg BID plus E2/NETA. AEs and SAEs during the Double-Blind treatment period were collected from the first dose of study drug to the start of the open label period (12 months).
- Open Label Placebo to Elagolix E2/NETA: For months 13 through 48, participants randomized to placebo in the 12-month double-blind treatment period switched to elagolix 300 mg BID plus E2/NETA during the open label treatment period. AEs and SAEs during the open label treatment period were collected from the first dose of open label study drug to the end of treatment.
- Open Label Elagolix E2 NETA to Elagolix E2/NETA: For months 13 through 48, participants randomized to Double-Blind Elagolix E2/NETA in the 12-month double-blind treatment period continued receiving elagolix 300 mg BID plus E2/NETA during the open label treatment period. AEs and SAEs during the open label treatment period were collected from the first dose of open label study drug to the end of treatment.
- Follow-up: Placebo to Elagolix E2/NETA; Follow-up: Elagolix E2 NETA to Elagolix E2/NETA: Participants entered the 12-month PTFU period after the last dose of study drug (after completing treatment month 48 or at any time a participant prematurely discontinued during the treatment period). AEs and SAEs were collected from the end of treatment through the end of the PTFU period. Safety reporting during the PTFU period included Adverse Events of Special Interest (AESIs). Other AEs may have also been reported.
Arm/Group | Screening Placebo | Screening Elagolix E2/NETA | Double-Blind Placebo | Double-Blind Elagolix E2/NETA | Open Label Placebo to Elagolix E2/NETA | Open Label Elagolix E2 NETA to Elagolix E2/NETA | Follow-up: Placebo to Elagolix E2/NETA | Follow-up: Elagolix E2 NETA to Elagolix E2/NETA
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/319 | 0/159 | 1/319 | 0/84 | 0/193 | 0/159 | 1/319
Serious Adverse Events (participants affected / at risk) | 1/159 | 3/319 | 2/159 | 10/319 | 7/84 | 9/193 | 1/159 | 3/319
Other Adverse Events (participants affected / at risk) | 1/159 | 0/319 | 28/159 | 88/319 | 41/84 | 65/193 | 3/159 | 5/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Placebo (N=159) | Screening Elagolix E2/NETA (N=319) | Double-Blind Placebo (N=159) | Double-Blind Elagolix E2/NETA (N=319) | Open Label Placebo to Elagolix E2/NETA (N=84) | Open Label Elagolix E2 NETA to Elagolix E2/NETA (N=193) | Follow-up: Placebo to Elagolix E2/NETA (N=159) | Follow-up: Elagolix E2 NETA to Elagolix E2/NETA (N=319)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THYROID MASS (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROLAPSE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Placebo (N=159) | Screening Elagolix E2/NETA (N=319) | Double-Blind Placebo (N=159) | Double-Blind Elagolix E2/NETA (N=319) | Open Label Placebo to Elagolix E2/NETA (N=84) | Open Label Elagolix E2 NETA to Elagolix E2/NETA (N=193) | Follow-up: Placebo to Elagolix E2/NETA (N=159) | Follow-up: Elagolix E2 NETA to Elagolix E2/NETA (N=319)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 11 (12) | 24 (27) | 0 (0) | 0 (0)
TRICHOMONIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
BONE DENSITY DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 16 (16) | 8 (8) | 27 (27) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 9 (10) | 6 (8) | 4 (4) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (9) | 12 (12) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 17 (19) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 4 (5) | 6 (6) | 7 (7) | 3 (3) | 0 (0) | 2 (2)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 4 (5) | 11 (18) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 6 (6) | 30 (34) | 6 (6) | 3 (3) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 9 (9) | 5 (5) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT03271489/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03271489/SAP_001.pdf